CLINICAL TRIAL: NCT01693029
Title: Randomized, Double-blind, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of HX575 Epoetin Alfa vs. US Licensed Epoetin Alfa (Epogen®/Procrit®) in the Treatment of Anemia Associated With Chronic Kidney Disease
Brief Title: Study to Compare Safety and Efficacy of HX575 Epoetin Alfa and US-licensed Epoetin Alfa
Acronym: ACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX575-307
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Anemia; Chronic Kidney Disease (CKD)
Keywords: erythropoietin alfa; CKD 5d
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HX575 epoetin alfa (Experimental): HX575, recombinant human epoetin alfa
  Interventions: Drug: HX575 epoetin alfa
- US-licensed epoetin alfa (Active Comparator): US-licensed recombinant human epoetin alfa
  Interventions: Drug: US-licensed epoetin alfa

INTERVENTIONS:
Drug: HX575 epoetin alfa — Solution for subcutaneous injection. The drug is administered subcutaneously at least once per week over 52 weeks. The dose will be individually titrated to maintain hemoglobin levels between 10 to 11 g/dL.
  Other Names: Binocrit® (Europe); Epoetin alfa HEXAL® (Europe); Abseamed® (Europe)
  Arms: HX575 epoetin alfa
Drug: US-licensed epoetin alfa — Solution for subcutaneous injection.
  Other Names: Epogen®; Procrit®
  Arms: US-licensed epoetin alfa

SUMMARY:
The purpose of this study is to show biosimilarity of HX575 epoetin alfa with the US licensed reference product Epogen®/Procrit® when applied subcutaneously. This study is intended to generate data supporting that the efficacy and safety under treatment with HX575 and Epogen®/Procrit® are comparable.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, multicenter study to evaluate the efficacy and safety of HX575 epoetin alfa vs. US-licensed epoetin alfa (Epogen®/Procrit®) in the treatment of anemia associated with chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease (stage CKD 5d), receiving stable subcutaneous maintenance therapy with Epogen® or Procrit® at least once per week
* Mean hemoglobin level between 9.0 - 11.5 g/dL during the screening period
* Adequate iron substitution

Exclusion Criteria:

* Contraindications for Erythropoiesis Stimulating Agent (ESA) therapy
* History of Pure Red Cell Aplasia (PRCA), or anti-erythropoietin (EPO) antibodies
* Known Human Immunodeficiency Virus (HIV) or Hepatitis B infection
* Hepatitis C infection on an active treatment
* Symptomatic congestive heart failure (New York Heart Association [NYHA] class III and IV)
* Unstable angina pectoris, or cardiac infarction during the last 6 months prior to randomization
* Percutaneous coronary intervention, or coronary artery bypass grafting during the last 6 months prior to randomization
* History of malignancy of any organ system
* Systemic lupus erythematous
* Immunocompromized patients

Other In-/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceutical Clinical Development, Study Director — Sandoz Biopharmaceuticals
Locations (52):
- United States (52):
  - Southwestern Kidney Institute, Tempe, Arizona
  - North America Research Institute, Azusa, California
  - Pegasus Dialysis, LLC, Bakersfield, California
  - Central Nephrology Medical Group, Bakersfield, California
  - California Institute of Renal Research, Chula Vista, California
  - Renal Consultants Medical Group, Granada Hills, California
  - Angel Kidney Care of Inglewood Dialysis Center, Inglewood, California
  - California Institute of Renal Research, La Mesa, California
  - Alliance Research Centers, Laguna Hills, California
  - Academic Medical Research Institute, Los Angeles, California
  - Ronald Reagan Medical Center, Department of Pharmaceutical Services, Drug Information Center, Los Angeles, California
  - Tower Nephrology Medical Group, Los Angeles, California
  - St Vincent Dialysis Center, Los Angeles, California
  - Kidney Research Center, Lynwood, California
  - Valley Renal Medical Group, Northridge, California
  - Ontario Dialysis, Inc., Ontario, California
  - Apex Research of Riverside, Riverside, California
  - Capital Nephrology Medical Group, Sacramento, California
  - California Institute of Renal Research, San Diego, California
  - La Jolla Clinical Research, Inc., San Diego, California
  - North America Research Institute, San Dimas, California
  - American Institute of Research, Whittier, California
  - South Florida Nephrology, Coral Springs, Florida
  - Pines Clinical Research Inc., Hollywood, Florida
  - Genesis Clinical Research Corporation, Tampa, Florida
  - Atekha Nephrology Clinic LLC, Statesboro, Georgia
  - Four Rivers Clinical Research, Incorporated, Paducah, Kentucky
  - Northwest Louisana Nephrology, Shreveport, Louisiana
  - Germantown Dialysis, Germantown, Maryland
  - Fresenius Management Services, Inc., Farmington, Missouri
  - Creighton University, Omaha, Nebraska
  - Kidney Specialists of Southern Nevada, Las Vegas, Nevada
  - Seacoast Kidney and Hypertension Specialist, PLLC, Portsmouth, New Hampshire
  - Renal Medicine Associates, Albuquerque, New Mexico
  - New York Hospital Queens, Fresh Meadows, New York
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Boice-Willis Clinic, PA, Rocky Mount, North Carolina
  - Southeastern Dialysis Center, Wilmington, North Carolina
  - Northeast Clinical Research Centers, Inc., Bethlehem, Pennsylvania
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Nephrology PA, Orangeburg, South Carolina
  - SC Nephrology & Hypertension Center, Inc., Orangeburg, South Carolina
  - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - Research Management, Inc., Austin, Texas
  - Gamma Clinical Research Institute, Edinburg, Texas
  - Nephrology, P.A., Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Renal Associates, PA, San Antonio, Texas
  - Southern Utah Kidney and Hypertension Center, St. George, Utah
  - Mendez Center For Clinical Research, LLC, Alexandria, Virginia
  - West Virginia University Hospitals and Clinic, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Weir MR, Pergola PE, Agarwal R, Fink JC, Kopyt NP, Singh AK, Kumar J, Schmitt S, Schaffar G, Rudy A, McKay JP, Kanceva R. A Comparison of the Safety and Efficacy of HX575 (Epoetin Alfa Proposed Biosimilar) with Epoetin Alfa in Patients with End-Stage Renal Disease. Am J Nephrol. 2017;46(5):364-370. doi: 10.1159/000481736. Epub 2017 Oct 30. PMID 29084409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
Started (437 patients were randomized but 2 were excluded from analyses due to improper ICF signature process) | 217 | 218
Completed | 173 | 161
Not Completed | 44 | 57
Not completed — Withdrawal by Subject | 15 | 22
Not completed — Kidney transplantation | 7 | 7
Not completed — Bindinging anti-EPO antibodies | 6 | 2
Not completed — Protocol Violation | 6 | 7
Not completed — Change in dialysis modality | 2 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 6
Not completed — Death | 5 | 8
Not completed — Non-compliance | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa | Total
Number analyzed (Participants) | 217 | 218 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (13.76) | 57.6 (13.40) | 58.7 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 103 | 185
  Male | 135 | 115 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 93 | 188
  Not Hispanic or Latino | 122 | 125 | 247
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 5 | 16
  Asian | 6 | 13 | 19
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 57 | 72 | 129
  White | 139 | 128 | 267
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 217 | 218 | 435
Height [Mean (Standard Deviation); unit: cm] | 167.2 (10.17) | 166.0 (10.33) | 166.6 (10.26)
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (20.75) | 86.5 (24.32) | 84.6 (22.66)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.55 (6.872) | 31.41 (8.783) | 30.48 (7.933)
Primary cause of Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants]
  Diabetes mellitus | 115 | 122 | 237
  Hypertension | 65 | 52 | 117
  Chronic glomerulonephritis | 13 | 16 | 29
  Kidney abnormalities | 8 | 11 | 19
  Polycystic kidney disease | 5 | 4 | 9
  Urinary tract obstruction | 2 | 0 | 2
  Vasculitis | 2 | 0 | 2
  Amyloidosis | 1 | 0 | 1
  Unknown | 3 | 9 | 12
  Other | 3 | 4 | 7
Type of last Erythropoiesis Stimulating Agent (ESA) therapy prior [Count of Participants; unit: Participants]
  Epogen | 217 | 215 | 432
  Procrit | 0 | 3 | 3
Time since start of ESA therapy [Median (Inter-Quartile Range); unit: months] | 30.59 [13.01 to 54.01] | 36.24 [17.15 to 62.09] | 32.95 [14.85 to 59.20]
Time since start of dialysis [Median (Inter-Quartile Range); unit: months] | 36.11 [18.53 to 66.40] | 41.08 [22.54 to 63.64] | 38.60 [20.93 to 64.23]
Method of dialysis at Baseline [Count of Participants; unit: Participants]
  Hemodialysis | 192 | 192 | 384
  Peritoneal dialysis | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Hemoglobin Levels Between the Screening/Baseline Period (Week -4 to Day 1) and the Evaluation Period (Week 21-28)
Description: Response to epoetin alfa in anemic patients with chronic renal failure is manifested by increased hematocrit, hemoglobin, reduced transfusion requirements and increase in quality of life. Hemoglobin (laboratory haematology parameter) is the primary endpoint of the study .
Time Frame: Week -4 to Day1 and Week 21-28
Population: The intent-to-treat (ITT) population consists of all randomized patients who were exposed to treatment with study drug for at least four weeks and have at least one Hb value available at week 4 or later. Following the intent-to-treat principle, patients are analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
Number analyzed (Participants) | 210 | 212
g/dL | -0.0960 (0.0575) | -0.0035 (0.0573)
Statistical Analysis 1: Comparison: HX575 Epoetin Alfa vs US-licensed Epoetin Alfa; Test type: Equivalence — Equivalence margin (-0.5, 0.5) g/dL. Results from ANCOVA with factors "treatment group" and covariates mean baseline Hb and mean weekly dose during the evaluation period (Week 21-28); Mean Difference (Final Values) = -0.0926, 90% CI 2-sided [-0.2264 to 0.0413]; 95% confidence interval for the difference is (-0.2522, 0.0670)

2. Primary Outcome: Change in Mean Hb Level Between Baseline (Week -4 to Day1) and Evaluation Period (Week 21-28)
Description: as for outcome 1
Time Frame: Week -4 to Day1 and Week 21-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
Number analyzed (Participants) | 210 | 212
g/dL
  Baseline period | 10.53 (0.635) | 10.50 (0.615)
  Evaluation period | 10.42 (0.826) | 10.51 (0.873)
  Change from baseline period to evaluation period | -0.11 (1.011) | 0.01 (0.953)

3. Secondary Outcome: Mean Weekly Dose During Evaluation Period (Week 21-28)
Description: Mean weekly study drug dose during evaluation period (Week 21-28)
Time Frame: Week 21-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: international units
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
Number analyzed (Participants) | 210 | 212
international units | 5876.5 (5785.50) | 5804.0 (6343.70)

4. Secondary Outcome: Incidence of Antibody Formation Against Epoetin
Description: Number of patients with positive antidrug antibody (ADA) finding at any time during their treatment period. Count includes 2 patients (1 in each arm) that already had a positive ADA Baseline finding. ADA testing performed by by Radio-Immuno-Precipitation assay. No patient developed neutralizing antibodies.
Time Frame: 52 weeks
Population: All patients treated with study drug with a post-baseline antibody assessment
Measure: Count of Participants; unit: Participants
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
Number analyzed (Participants) | 214 | 216
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of informed consent until the end of the treatment period, for approximately 1 year.
Description: Adverse events recorded before first study drug were considered pre-treatment adverse events, adverse events recorded more than 30 days after last study drug treatment were considered post-treatment emergent adverse event. Only treatment-emergent adverse events are shown in adverse events counts.
Arm/Group | HX575 Epoetin Alfa | US-licensed Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 5/217 | 11/218
Serious Adverse Events (participants affected / at risk) | 91/217 | 90/218
Other Adverse Events (participants affected / at risk) | 112/217 | 123/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa (N=217) | US-licensed Epoetin Alfa (N=218)
Pneumonia (Infections and infestations) | 9 (9) | 10 (12)
Cellulitis (Infections and infestations) | 7 (8) | 7 (7)
Peritonitis (Infections and infestations) | 5 (6) | 3 (3)
Gangrene (Infections and infestations) | 3 (3) | 4 (7)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Staphylococcal bacteraemia (Infections and infestations) | 5 | 5 (5)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 | 2 (3)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 0
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 | 2 (2)
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 (2)
Abscess neck (Infections and infestations) | 1 (1) | 0
Diverticulitis (Infections and infestations) | 1 (1) | 0
Intervertebral discitis (Infections and infestations) | 1 (1) | 0
Staphylococcal infection (Infections and infestations) | 1 (1) | 0
Urosepsis (Infections and infestations) | 1 (1) | 0
Abdominal abscess (Infections and infestations) | 0 | 1 (1)
Catheter site infection (Infections and infestations) | 0 | 1 (1)
Device related sepsis (Infections and infestations) | 0 | 1 (1)
Endocarditis (Infections and infestations) | 0 | 1 (1)
Gastroenteritis (Infections and infestations) | 0 | 1 (1)
Influenza (Infections and infestations) | 0 | 1 (1)
Salmonellosis (Infections and infestations) | 0 | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 (1)
Viral infection (Infections and infestations) | 0 | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 8 (9) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 7 (8)
Cardiac arrest (Cardiac disorders) | 4 (4) | 3 (4)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2)
Coronary artery disease (Cardiac disorders) | 5 (5) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0
Myocardial infarction (Cardiac disorders) | 1 (1) | 0
Palpitations (Cardiac disorders) | 1 (1) | 0
Cardiovascular deconditioning (Cardiac disorders) | 0 | 1 (1)
Tachycardia (Cardiac disorders) | 0 | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (9) | 7 (8)
Fluid overload (Metabolism and nutrition disorders) | 6 (6) | 8 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4 (4)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 2 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 (2)
Colitis (Gastrointestinal disorders) | 0 | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 0 | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 4 (5)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (7) | 2 (2)
Medical device complication (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 0
Asthenia (General disorders) | 0 | 3 (3)
Device malfunction (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 | 2 (2)
Catheter site pain (General disorders) | 0 | 1 (2)
Chest pain (Injury, poisoning and procedural complications) | 1 (1) | 0
Necrosis (General disorders) | 1 (1) | 0
Pain (General disorders) | 1 (1) | 0
Chest discomfort (General disorders) | 0 | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 4 (5)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 | 2 (2)
Malignant hypertension (Vascular disorders) | 1 (1) | 0
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0
Accelerated hypertension (Vascular disorders) | 0 | 1 (1)
Lymphoedema (Vascular disorders) | 0 | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0
Encephalopathy (Nervous system disorders) | 1 (1) | 0
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0
Myoclonus (Nervous system disorders) | 1 (1) | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 | 1 (1)
Presyncope (Nervous system disorders) | 0 | 1 (1)
Speech disorder (Nervous system disorders) | 0 | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0
Mental status changes (Psychiatric disorders) | 1 (1) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0
Renal mass (Renal and urinary disorders) | 1 (1) | 0
Urinary retention (Renal and urinary disorders) | 1 (1) | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 (2)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0
Biliary tract dilation procedure (Surgical and medical procedures) | 1 (1) | 0
Troponin increased (Investigations) | 0 | 1 (1)
Treatment noncompliance (Social circumstances) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa (N=217) | US-licensed Epoetin Alfa (N=218)
Upper respiratory tract infection (Infections and infestations) | 12 (14) | 22 (24)
Urinary tract infection (Infections and infestations) | 12 (15) | 10 (13)
Fall (Injury, poisoning and procedural complications) | 13 (20) | 18 (31)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 15 (17) | 11 (16)
Diarrhoea (Gastrointestinal disorders) | 21 (26) | 19 (24)
Nausea (Gastrointestinal disorders) | 17 (20) | 20 (23)
Vomiting (Gastrointestinal disorders) | 10 (18) | 15 (18)
Constipation (Gastrointestinal disorders) | 10 (10) | 13 (13)
Pyrexia (General disorders) | 12 (16) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16) | 16 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 14 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (13) | 14 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (11) | 11 (12)
Hypertension (Vascular disorders) | 24 (40) | 27 (34)
Hypotension (Vascular disorders) | 9 (10) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 15 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (12)
Headache (Nervous system disorders) | 15 (17) | 15 (18)
Dizziness (Nervous system disorders) | 9 (11) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.